CLINICAL TRIAL: NCT02074111
Title: Moyamoya Disease Biomarkers in Patients With Intracranial Atherosclerotic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Oh Young Bang, Associate Professor, Samsung Medical Center
Other Study IDs: 2013-08-098-003
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Moyamoya Disease; Intracranial Atherosclerotic Stroke; Intracranial Steno-occlusive Disease
Keywords: Moyamoya disease; Intracranial atherosclerotic stroke; Intracranial steno-occlusive disease; ring finger 213 (RNF213) gene mutation; high-resolution MRI
MeSH Terms: conditions — Moyamoya Disease; Moyamoya disease 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Intracranial atherosclerotic stroke
- Moyamoya disease
- Healthy controls

SUMMARY:
The aim of this study is to investigate the proportion of patients with moyamoya disease among the patients who were diagnosed as having intracranial atherosclerotic stroke. To do this, biomarkers (gene and imaging) for moyamoya disease are tested and follow up angiography are performed during follow up (in selected patients).

DETAILED DESCRIPTION:
1. Purpose Both moyamoya disease (MMD) and intracranial atherosclerotic stenosis (ICAS) are more prevalent in Asians than in Westerners, although the reason for the race-ethnic differences is unsettled. It is possible that patients with adult-onset MMD were misclassified as having ICAS, which may in part explain the high prevalence of intracranial atherosclerosis in Asians. It is important to differentiation between these two diseases because MMD and ICAS have differential therapeutic strategies (surgical revascularization in MMD vs. the use of antithrombotics/statins and stenting in ICAS). The ring finger 213 (RNF213) was recently identified as a susceptibility gene for MMD in East Asians. Characteristic high-resolution (HR) MRI findings of MMD and ICAS have recently been reported. The aim of this study is to investigate the proportion of patients with moyamoya disease among the patients who were diagnosed as having intracranial atherosclerotic stroke. To do this, biomarkers (gene and imaging) for moyamoya disease are tested and follow up angiography are performed during follow up (in selected patients).
2. Conditions: Stroke, intracranial occlusive lesion
3. Intervention: None
4. Study period: Jan 22, 2014 ~ Dec 31, 2016
5. Study design: Observational model Time perspective: Retrospective-Prospective

ELIGIBILITY:
Inclusion Criteria:

1. Intracranial atherosclerotic stroke

   * Patients with age over 20 years
   * Patients with focal neurological deficits presented within 7 days of symptom onset
   * Patients with acute ischemic lesions on diffusion-weighted image (DWI)
   * Patients with stenosis on the relevant intracranial vessels (distal ICA and/ or M1)
2. Moyamoya disease

   * Patients with age over 20 years
   * Patients who performed conventional angiography
   * Patients who are diagnosed as having either definite or probable Moyamoya disease
3. Healthy subjects

   * Subjects with age over 20 years
   * Subjects with no history of cerebrovascular disease

Exclusion Criteria:

* Patients with extracranial stenosis more than 50%
* Patients with potential sources of cardio-aortic embolism
* Patients with moderate to severe renal disease
* Pregnancy or lactation
* Patients with short life expectancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tertiary Hospital
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of RNF213 gene variants and HR-MRI findings in patients with intracranial atherosclerosis | Anytime during study period (in intracranial atherosclerosis, HR-MRI findings within 2 weeks)

SECONDARY OUTCOMES:
Frequency of typical angiographic findings of moyamoya disease at follow up conventional angiography in patients with intracranial atherosclerosis who showed typical gene and imaging biomarkers of moyamoya disease | Within 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Oh Young Bang, MD PhD, Principal Investigator — Associate Professor
Locations (1):
- Department of Neurology, Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim JY, Kim HJ, Choi EH, Pan KH, Chung JW, Seo WK, Kim GM, Jee TK, Yeon JY, Kim JS, Hong SC, Seong MJ, Cha J, Kim KH, Jeon P, Bang OY. Vessel Wall Changes on Serial High-Resolution MRI and the Use of Cilostazol in Patients With Adult-Onset Moyamoya Disease. J Clin Neurol. 2022 Nov;18(6):610-618. doi: 10.3988/jcn.2022.18.6.610. PMID 36367058